CLINICAL TRIAL: NCT04303611
Title: To Examine the Role of Family Support for Patients With Obesity Before and After Bariatric Surgery and Whether Family Support Predicts Long-term Weight Loss and Diabetes Outcomes
Brief Title: Examining The Role of Family Support in Bariatric Surgery Patients
Status: Completed | Type: Observational
Sponsor: Yale-NUS College (Other)
Responsible Party: Sponsor
Other Study IDs: 9737926B
Record Dates: First submitted 2020-03-08; First posted 2020-03-11 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2018-10

CONDITIONS: Focus of Study is Patient Responses to an Obesity Management Questionnaire Administered by SGH Life Centre

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to examine the role of family support on the adhesion to post-op procedures in patients who have undergone bariatric surgery in Singapore.

ELIGIBILITY:
Inclusion Criteria:

Undergone bariatric surgery within SGH Life Centre and must have completed the intake questionnaire

Exclusion Criteria:

-

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Undergone bariatric surgery within SGH Life Centre and completed the intake questionnaire
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2018-08-13 (Actual); Primary Completion 2018-09-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Weight Loss | Immediately post-surgery within first year
  Weight Loss in Kilograms

CONTACTS AND LOCATIONS:
Locations (1):
- Singapore General Hospital, Singapore, Singapore

REFERENCES:
- [Derived] Tan EY, Lee PC, Tham KW, Ganguly S, Lim CH, Liu JCJ. Examining spousal and family support as predictors of long-term weight loss and remission of type 2 diabetes following bariatric surgery in Singapore: a retrospective cohort study. BMJ Open. 2023 May 2;13(5):e068810. doi: 10.1136/bmjopen-2022-068810. PMID 37130681